CLINICAL TRIAL: NCT05543005
Title: Efficacy Study of an Audio Device Outside Incubator Allowing Broadcasting Maternal Voice on Stability in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia-Jung Lin (Other)
Responsible Party: Sponsor-Investigator, Chia-Jung Lin, nurse practitioner, Far Eastern Memorial Hospital
Organization: Far Eastern Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 111119-F
Record Dates: First submitted 2022-08-30; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Premature Infant
Keywords: premature infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The study designs a two-arm, double blind randomized control trial (RCT) experiment in terms of a block randomization for allocating participants in experimental and control groups respectively. In the experimental group maternal voice in terms of lullaby, music, and meaningful words plays near the head of premature infant in the incubator by 30 mins each time, and totally three times a day over a 14-days intervention duration. Meanwhile a standard care treats premature infants in the control group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): maternal voice
  Interventions: Other: maternal voice intervention
- control group (No Intervention): no maternal voice

INTERVENTIONS:
Other: maternal voice intervention — maternal voice in terms of lullaby, music, and meaningful words plays near the head of premature infant in the incubator by 30 mins each time after routine care period
  Arms: experimental group

SUMMARY:
The study aims to evaluate the impact on the preterm infants' short-term physiological, neurodevelopmental states by employing maternal voice intervention in NICU routine care. This study also evaluates the correlation between effective intervention and maternal depression by employing Edinburgh Postnatal Depression Scale .

DETAILED DESCRIPTION:
The study designs a two-arm, double blind randomized control trial (RCT) experiment in terms of a block randomization for allocating participants in experimental and control groups respectively. In the experimental group maternal voice in terms of lullaby, music, and meaningful words plays near the head of premature infant in the incubator by 30 mins each time, and totally three times a day over a 14-days intervention duration. Meanwhile a standard care treats premature infants in the control group. A IntelliVue physiological monitor and a behavior scale collects ECG, respiratory rate, SpO2 concentration, and sleep/awake states of premature infants in both groups. Finally, ANOVA analyzes the statistical significance between the measurer and items.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants at 28-36 gestational age
* Within 10 days in NICU after delivery

Exclusion Criteria:

1. Has a known chromosomal or congenital abnormality
2. Major congenital infection
3. Brain lesions diagnosed prenatally, or neonatal asphyxia at birth.
4. Toxic use by the mother during pregnancy
5. Intraventricular hemorrhage of third degree or more occurred in brain ultrasound examination
6. Are using sedative medication
7. Premature infants use endotracheal tube respirator or high-frequency respirator
8. Preterm infants requiring immediate surgical treatment at birth

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
heart rate | 14th day
  observation at 7th and 14th day after intervention period
respiratory rate | 14th day
  observation at 7th and 14th day after intervention period
SpO2 concentration | 14th day
  observation at 7th and 14th day after intervention period
behavioral status with crying states of premature infants | 14th day
  observation at 7th and 14th day after intervention period